CLINICAL TRIAL: NCT01808898
Title: Randomized Double-blind Placebo Controlled Trial to Assess the Role of Intrauterine Cornual Block (ICOB) in Combination With Direct Cervical Block in Outpatient Endometrial Ablation
Brief Title: Role of Intrauterine Cornual Block in Combination With Direct Cervical Block in Outpatient Endometrial Ablation
Acronym: ICOB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 12/BWH/NO75
Record Dates: First submitted 2013-02-24; First posted 2013-03-11 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2015-05

CONDITIONS: Endometrial Diseases
Keywords: Ablation; Outpatient
MeSH Terms: conditions — Uterine Diseases | interventions — Anesthesia, Local; Mepivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local anaesthetic (Experimental): 2mls consisting of 1ml of 3% mepivacaine (short / medium acting) and 1ml of 0.5% bupivacaine (long acting)
  Interventions: Procedure: Local Anaesthetic
- Saline (Placebo Comparator): 2mls of Normal Saline solution in a 5ml syringe
  Interventions: Procedure: Local Anaesthetic

INTERVENTIONS:
Procedure: Local Anaesthetic — On the day of the procedure and before the patients are treated, a designated clinician will draw up the local anaesthetic (2mls consisting of 1ml of 3% mepivacaine (short / medium acting) and 1ml of 0.5% bupivacaine (long acting)
  Other Names: Mepivacaine and bupivacaine

SUMMARY:
The usual intervention to control the pain during an outpatient endometrial ablation has been to use local anaesthesia (LA) injection just in the neck of the womb (cervix). However, this alone may not be sufficient to control the pain completely. Therefore, we want to find out whether an injection of LA given deep into the muscle of the womb (myometrium), in addition to that in the cervix, has a better effect on controlling the pain during the procedure.

All women attending gynaecology outpatient clinics, who have consented for an outpatient hysteroscopic procedure, will be invited to take part in the study. The study will be carried out in the outpatient hysteroscopy clinic at Birmingham Women's Hospital.

As part of standard pain control method during an outpatient endometrial ablation, all women will receive an injection of LA in the cervix of the uterus to 'freeze it'. During hysteroscopy a randomly selected treatment group will receive an injection into deep muscle containing only normal saline (control group) whereas the experiment group will receive fast / long acting local anaesthesia (cornual block).

Women will be asked to rate the degree of pain by placing a mark on an ungraduated 10 cm horizontal line. These scales will be given before the procedure, during LA injection, immediately after, one hour and at the time of discharge from hospital.

The results will help future patients undergoing a similar procedure to have much better pain relief and allow many more to have the procedure without the side effects of a general anaesthetic and its risks. In addition to having less pain, it may reduce the number of painkillers needed as well as any stay in hospital. In future this may also allow a greater variety of procedures to be done in an outpatient setting.

DETAILED DESCRIPTION:
Outpatient local anaesthesic (LA) hysteroscopic intrauterine therapeutic interventions such as endometrial ablation have gained wider acceptance in the last decade. However, pain experienced during these procedures can be a disincentive and is the commonest reason for the use of escalating levels of analgesia post procedure, which results in prolongation of hospital stay and recovery. Various methods of LA have been studied including intrauterine topical lignocaine or cervical block using topical lignocaine, paracervical block or intracervical block. However, a single site block individually may not be sufficient to control the pain completely due to inability of the one site block to affect the sensitivity of the whole uterus, as the uterine fundus is effectively still unanaesthetised. This may be due to the uterus receiving complex innervations from different nerve routes such as the uterovaginal plexus, the Frankenhauser nerve plexuses, parasympathetic ganglia and the thoracic nerve.

Therefore, it seems logical to use a direct cervical block to block the sensation through uterovaginal plexus and use an additional deep myometrial block adjacent to each cornua to directly block the thoracic nerve supply. To date, only one small observational study has looked at the effect of such a combined block in relieving pain during outpatient hysteroscopic procedures. Therefore, we propose to undertake a double blind randomised controlled trial to address this question by comparing effectiveness of a standard direct cervical block and intrauterine cornual block (ICOB) versus a direct cervical block and a normal saline intrauterine cornual injection (control).

ELIGIBILITY:
Inclusion Criteria:

* All women between the ages of 18 - 50 years presenting to the gynaecology outpatient clinic scheduled for an outpatient hysteroscopic intrauterine therapeutic intervention such as endometrial ablation.

Exclusion Criteria:

* Women with contraindications to hysteroscopic procedures such as atypical endometrial hyperplasia or endometrial cancer, undiagnosed abnormal vaginal bleeding, current lower pelvic infection or uterine abnormalities

  * Women who are allergic to local anaesthesia
  * Not technically possible to perform a hysteroscopy e.g. women with distorted uterine cavity due to large fibroids
  * Women considered vulnerable (e.g. current mental illness, emotionally labile, or learning difficulties)
  * Women who decline to be randomised and request the additional anaesthetic or decline it will form a separate group to be studied and will be administered the VAS similar to the trial group. This group will be analysed separately to determine whether they are significantly different to those patients who consent to being part of the trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale evaluating pain | administered immediately after the procedure
  To determine the effectiveness of intrauterine cornual block by evaluating pain directly attributable to outpatient hysteroscopic endometrial ablation assessed by using an ungraduated 10 cm visual analogue scale (VAS) administered immediately after the procedure prior to shifting patient to the recovery unit.

SECONDARY OUTCOMES:
Visual Analogue scale evaluating pain | 1 hour after procedure and at discharge from hospital
  1. To determine the effectiveness of intrauterine cornual block by evaluating pain using VAS at 1 hour after the procedure and prior to discharge from the hospital.
  2. To assess the total requirements for rescue analgesia in the first 24-hour post-operative period between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Janesh K Gupta, MSc MD FRCOG, Principal Investigator — Birmingham University
Locations (1):
- Birmingham Women's Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Kumar V, Tryposkiadis K, Gupta JK. Hysteroscopic local anesthetic intrauterine cornual block in office endometrial ablation: a randomized controlled trial. Fertil Steril. 2016 Feb;105(2):474-80.e1. doi: 10.1016/j.fertnstert.2015.10.019. Epub 2015 Nov 4. PMID 26546298